CLINICAL TRIAL: NCT04484870
Title: Comparative Study on the Efficacy of Danshu Capsule and Ursodeoxycholic Acid Capsule in Preventing Recurrence of Choledocholithiasis
Brief Title: Danshu Capsule and Ursodeoxycholic Acid Capsule in Preventing Recurrence of Choledocholithiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, ZhangXiaofeng, Director of Department of Gastroenterology, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: （109）-1
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Choledocholithiasis; Recurrence
MeSH Terms: conditions — Choledocholithiasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danshu capsule group (Experimental): The patients in Danshu group were treated with Danshu capsule, 2 tablets per time, 3 times a day (0.45g/ tablets)，The course of treatment was 6 months
  Interventions: Drug: oral Danshu capsule
- ursodeoxycholic acid group (Active Comparator): UDCA group, 250mg/ was taken orally twice a day (0.25g/, Losan Pharma GmbH company). The course of treatment was 6 months
  Interventions: Drug: oral Danshu capsule

INTERVENTIONS:
Drug: oral Danshu capsule — Danshu group oral Danshu capsule, 2 tablets per time, 3 times a day (0.45g/ tablets, Sichuan Jishengtang Pharmaceutical Co., Ltd.)

SUMMARY:
[objective] to compare the efficacy of Danshu capsule and ursodeoxycholic acid (UDCA) in preventing recurrence of choledocholithiasis after operation. [methods] one hundred and fifty ERCP patients with choledocholithiasis were randomly divided into two groups: Danshu group (n = 75) and UDCA group (n = 75). The Danshu group took 2 Danshu capsules three times a day, and the UDCA group took 250 mg of Ursofalk twice a day. The clinical efficacy, changes of liver function indexes before and after treatment and stone recurrence were compared between the two groups.

ELIGIBILITY:
inclusion criteria:

1. Choledocholithiasis was diagnosed by B-ultrasound / CT/MRCP, The patients are generally in good condition, no surgical taboos, and can tolerate general anesthesia and ERCP surgery.
2. Agree to participate in the project research, know the benefits and possible risks of surgery, know the benefits and risks of drugs, and sign an informed consent form.

exclusion criteria：

1. patients with cholecystolithiasis, hepatitis B, biliary ascariasis, liver cirrhosis, hemolytic anemia, congenital jaundice and tumor were excluded.
2. Excluding serious primary diseases such as heart, brain, lung, kidney and blood system.
3. Those who are allergic or allergic to drugs in this test are excluded.
4. Pregnancy vibration or nursing women were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
recurrence rate | 1 year
  abdominal ultrasound or MRCP/CT was used to examine every 3 months after operation for 1 year, and the recurrence was recorded.

SECONDARY OUTCOMES:
improvement rate of liver function index | 3 days, 1 week and 2 weeks
  5ml of fasting elbow venous blood was taken before treatment and 3 days, 1 week and 2 weeks after treatment respectively. The blood samples were centrifuged and the supernatant was taken. Total bilirubin (total bilirubin, TBil), glutamic pyruvic transaminase (Alanine aminotransferase, ALT), glutamic oxaloacetic transaminase (Aspartate aminotransferase, AST) and γ-glutamyl transpeptidase (γ-glutamyl transpeptidase, GGT)) in blood samples were detected by automatic biochemical analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, Zhang, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou first people's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No